CLINICAL TRIAL: NCT01262898
Title: A Randomized, Double-Blind, Placebo-Controlled Multicenter Phase II Study to Evaluate the Safety and Efficacy and Dose Response of 28 Days of Once-Daily Dosing of the Oral Motilin Receptor Agonist GSK962040, in Type I and II Diabetic Male and Female Subjects With Gastroparesis
Brief Title: Dose Response of 28 Days of Dosing of GSK962040 in Type I and II Diabetic Male and Female Subjects With Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114479; 2010-023186-21 (EudraCT Number)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Gastroparesis
Keywords: tolerability; pharmacokinetics; 13 C oral breath test; Type I and II Diabetes mellitus; gastroparesis; gut motility; phase II; pharmacodynamics; repeat dose; gastric emptying; symptoms; GSK962040
MeSH Terms: conditions — Gastroparesis | interventions — N-(3-fluorophenyl)-1-((4-(((3S)-3-methyl-1-piperazinyl)methyl)phenyl)acetyl)-4-piperidinamine; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK962040 (10 mg) (Experimental): GSK962040 10 mg
  Interventions: Drug: GSK962040 (5 mg tablet)
- GSK962040 (50 mg) (Experimental): GSK962040 50 mg
  Interventions: Drug: GSK962040 (25 mg tablet)
- GSK962040 (125 mg) (Experimental): GSK962040 125 mg
  Interventions: Drug: GSK962040 (125 mg tablet)
- Placebo (Experimental): Placebo
  Interventions: Drug: GSK962040 (5 mg tablet); Drug: GSK962040 (25 mg tablet); Drug: GSK962040 (125 mg tablet); Drug: Placebo

INTERVENTIONS:
Drug: GSK962040 (5 mg tablet) — 5 mg tablet
  Arms: GSK962040 (10 mg); Placebo
Drug: GSK962040 (25 mg tablet) — 25 mg tablet
  Arms: GSK962040 (50 mg); Placebo
Drug: GSK962040 (125 mg tablet) — 125 mg tablet
  Arms: GSK962040 (125 mg); Placebo
Drug: Placebo — matching placebo tablet
  Arms: Placebo

SUMMARY:
GSK962040 is a novel small molecule motilin agonist. The Phase I studies (MOT107043 and MOT109681) demonstrated that single doses of GSK962040 up to 150 mg and repeat dosing of up to 125 mg/day for 14 days were well tolerated with adverse events not occurring in greater prevalence than placebo, and no significant abnormal vital sign, ECG, or clinical laboratory findings. Pharmacokinetic parameters were linear and approximately dose proportional over the range of doses administered. Single doses of 50 mg - 150 mg GSK962040 significantly increased the rate of gastric emptying up to 40% as measured by the 13C octanoic acid stable isotope breath test. A similar effect of 50 mg and 125 mg on gastric emptying was observed throughout repeated dosing to healthy volunteers for 14-days.

The aims of the present investigation (MOT114479) are to assess the pharmacodynamic effects (gastric emptying and symptoms), safety, tolerability, and pharmacokinetics of GSK962040 after 28 days of once-daily dosing in Type I and Type II diabetic subjects with gastroparesis. An additional aim is to characterize the dose/exposure - pharmacodynamic effect relationship.

ELIGIBILITY:
Inclusion Criteria:

* Type I or II Diabetes Mellitus (HbA1C < 10%)
* Male or female between 18 and 80 years of age, inclusive.
* Patient has gastroparesis at screening (gastric half-time of emptying > upper limit of normal as determined by 13C-oral breath test)
* Patient must have a > or = 3 month history of relevant symptoms of gastroparesis (e.g., chronic post-prandial fullness, early satiety, postprandial nausea), patients will have a mean of the daily scores over a minimum of 7 days indicating > or = mild (2) and < or = severe (4) post-prandial fullness assessed using the GCSI-DD during the screening period prior to randomization.
* A female patient is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/mL, or a value consistent with the local laboratory standard value, is confirmatory. OR Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female patients must agree to use contraception for at least 5 days following the last dose of study medication.
* Male patients must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication through at least 5 days after the last dose of study medication.
* BMI >18 and < or = 35.0 kg/m2 (inclusive).
* Patient has never had a gastrectomy, nor major gastric surgical procedure or any evidence of bowel obstruction or strictures within the previous 12 months
* Dosage of any concomitant medications has been stable for at least 3 weeks, except for routine adjustments in daily insulin treatments.
* Estimated (or measured) glomerular filtration rate > or = 30 mL/min.
* QTcB or QTcF < 450 msec or QTc < 480 msec in patients with Bundle Branch Block based on single or average QTc value of triplicate values obtained over a brief recording period.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin < or = 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Exclusion Criteria:

* Patient has acute severe gastroenteritis
* Patient has a gastric pacemaker
* Patient is on chronic parenteral feeding
* Patient has pronounced dehydration
* Recent (last 6 weeks) history of poor control of diabetes e.g. hypoglycaemia requiring medical intervention, diabetic ketoacidosis, admission for control diabetes or complications of diabetes
* Patient has evidence of severe cardiovascular autonomic neuropathy (e.g. history of recurrent syncope in the last 6 months)
* Patient has a history of eating disorders (anorexia nervosa, binge eating, bulimia)
* Use of medications potentially influencing upper gastrointestinal motility or appetite within one week of the study (e.g., prokinetic drugs, macrolide antibiotics (erythromycin), GLP-1 mimetics)
* Regular opiate use
* Use of prohibited medications listed in Section 9.2 within the restricted timeframe relative to the first dose of study medication.
* History or presence of clinically significant gastro-intestinal, hepatic or renal disease or other condition that would in the opinion of the investigator or medical monitor make the subject unsuitable for inclusion in this clinical study.
* The patient has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day time-period.
* Pregnant females as determined by positive serum or urine hCG test (from the first urine of the day) at screening or prior to dosing.
* Lactating females.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-05-03 (Actual); Primary Completion 2013-02-26 (Actual); Study Completion 2013-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (9):
  - GSK Investigational Site, Concord, California
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Chevy Chase, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- GSK Investigational Site, Randwick, New South Wales, Australia
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Thornhill, Ontario
  - GSK Investigational Site, Toronto, Ontario
- GSK Investigational Site, Uppsala, Sweden
- United Kingdom (4):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, London
  - GSK Investigational Site, Salford

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 80 participants were enrolled and randomized from 03 May 2011 to 26 Feb 2013. The study was conducted at 22 centers, 1 center in Australia, 1 center in Sweden, 2 centers in Belgium, 4 centers in Canada, 5 Centers in United Kingdom and 9 centers in United States.
Pre-assignment Details: Out of 80 participants randomized, 1 participant withdrew consent prior to dosing in GSK962040 50 milligram (mg) arm. Remaining 79 participants were included in "All subject population"
Groups:
- Placebo: Participants received placebo tablets matching to GSK962040 administered orally once daily for a period of 28 days.
- GSK962040 10 mg: Participants received GSK962040 10 mg tablets administered orally once daily for a period of 28 days.
- GSK962040 50 mg: Participants received GSK962040 50 mg tablets administered orally once daily for a period of 28 days.
- GSK962040 125 mg: Participants received GSK962040 125 mg tablets administered orally once daily for a period of 28 days.
Period: Overall Study
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Started | 21 | 18 | 18 | 22
Completed | 18 | 16 | 18 | 22
Not Completed | 3 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg | Total
Number analyzed (Participants) | 21 | 18 | 18 | 22 | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (14.23) | 54.0 (11.42) | 55.2 (12.17) | 51.4 (11.34) | 53.7 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 10 | 9 | 47
  Male | 7 | 4 | 8 | 13 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 1 | 3
  Black or African American | 2 | 2 | 0 | 0 | 4
  White | 19 | 15 | 17 | 20 | 71
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Gastric Half Emptying Time (GEt1/2)
Description: Gastric half emptying time is the time taken for half the contents of the stomach to empty. Gastric emptying was measured using the 13C-oral breath test, which is a tracer method that utilizes 13C, a non-radioactive isotope. Basal breath samples were obtained after an overnight fast or otherwise after 4 hours of fasting following a light meal. On Day 1 and Day 28, participants were then dosed with GSK962040 and additional breath test samples were taken prior to administration of a 13C-labelled test meal. The test meal was consumed approximately 80 minutes(min) later. After consumption of the test meal, breath samples were collected at pre-specified time points over an approximately 4 hour period following the test meal. For the duration of the breath test, no food or drink were allowed. The 13C breath content was determined by isotope ratio mass spectrometry. GE t1/2 was determined by using the cumulative percentage of the administered dose of 13C excreted in breath over 4 hours.
Time Frame: Screening2/Baseline (Day -30 to -1) , Day 1, and Day 28
Population: The 'All Subjects Population' compromised of all participants who received at least one dose of study medication. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Minutes
  Baseline | 131.2 (25.31) | 106.5 (23.42) | 118.2 (31.13) | 131.1 (32.66)
  Day 1: number analyzed (Participants) | 21 | 18 | 18 | 21
  Day 1 | 124.1 (39.25) | 106.6 (27.07) | 104.8 (21.61) | 99.4 (33.55)
  Day 28: number analyzed (Participants) | 18 | 16 | 18 | 22
  Day 28 | 111.8 (24.37) | 111.8 (32.23) | 107.9 (29.03) | 117.8 (44.20)
Statistical Analysis 1: Comparison: Placebo vs GSK962040 10 mg; GSK962040 10 mg versus Placebo Day 1; Test type: Superiority or Other; Mean Difference (Net) = -3.36, 95% CI 2-sided [-21.96 to 15.24], Standard Deviation 14.47 — The least square means were estimated using a mixed model fitting treatment, visit, treatment*visit and baseline gastric emptying half time as fixed effects, and participant as a random effect. Statistical analysis is reported using LS Means
Statistical Analysis 2: Comparison: Placebo vs GSK962040 50 mg; GSK962040 50 mg versus Placebo Day 1; Test type: Superiority or Other; Mean Difference (Net) = -11.81, 95% CI 2-sided [-30.01 to 6.40], Standard Deviation 14.47 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs GSK962040 125 mg; GSK962040 125 mg versus Placebo Day 1; Test type: Superiority or Other; Mean Difference (Net) = -25.65, 95% CI 2-sided [-42.99 to -8.32], Standard Deviation 14.47 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs GSK962040 10 mg; GSK962040 10 mg versus Placebo Day 28; Test type: Superiority or Other; Mean Difference (Net) = 14.74, 95% CI 2-sided [-5.06 to 34.53], Standard Deviation 14.47 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs GSK962040 50 mg; GSK962040 50 mg vs Placebo Day 28; Test type: Superiority or Other; Mean Difference (Net) = 4.22, 95% CI 2-sided [-14.64 to 23.08], Standard Deviation 14.47 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs GSK962040 125 mg; GSK962040 125 mg versus Placebo Day 28; Test type: Superiority or Other; Mean Difference (Net) = 6.65, 95% CI 2-sided [-11.18 to 24.47], Standard Deviation 14.47 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo; Day 28 versus Day 1 of the Placebo arm; Test type: Superiority or Other; Mean Difference (Net) = -12.92, 95% CI 2-sided [-28.73 to 2.90], Standard Deviation 14.47 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: GSK962040 10 mg; Day 28 versus Day 1 of GSK962040 10 mg arm; Test type: Superiority or Other; Mean Difference (Net) = 5.18, 95% CI 2-sided [-11.69 to 22.05], Standard Deviation 14.47 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: GSK962040 50 mg; Day 28 versus Day 1 of GSK962040 50 mg arm; Test type: Superiority or Other; Mean Difference (Net) = 3.11, 95% CI 2-sided [-13.13 to 19.36], Standard Deviation 14.47 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: GSK962040 125 mg; Day 28 versus Day 1 of GSK962040 125 mg arm; Test type: Superiority or Other; Mean Difference (Net) = 19.39, 95% CI 2-sided [4.47 to 34.30], Standard Deviation 14.47 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs GSK962040 10 mg vs GSK962040 50 mg vs GSK962040 125 mg; Type 1 Diabetes, Day 1; Test type: Superiority or Other; Mixed Models Analysis; Slope = -0.225, 95% CI 2-sided [-0.320 to -0.129]; Intercept estimate was 125.45 and between participant standard deviation was 21.63
Statistical Analysis 12: Comparison: Placebo vs GSK962040 10 mg vs GSK962040 50 mg vs GSK962040 125 mg; Type 1 Diabetes, Day 28; Test type: Superiority or Other; Mixed Models Analysis; Slope = -0.078, 95% CI 2-sided [-0.171 to 0.016]; Intercept estimate was 125.45 and between participant standard deviation was 21.63
Statistical Analysis 13: Comparison: Placebo vs GSK962040 10 mg vs GSK962040 50 mg vs GSK962040 125 mg; Type 2 Diabetes, Day 1; Test type: Superiority or Other; Mixed Models Analysis; Slope = -0.225, 95% CI 2-sided [-0.320 to -0.129]; Intercept estimate was 113.23 and between participant standard deviation was 21.63
Statistical Analysis 14: Comparison: Placebo vs GSK962040 10 mg vs GSK962040 50 mg vs GSK962040 125 mg; Type 2 Diabetes, Day 28; Test type: Superiority or Other; Mixed Models Analysis; Slope = -0.078, 95% CI [-0.171 to 0.016]; Intercept estimate was 113.23 and between participant standard deviation was 21.63

2. Secondary Outcome: Number of Participants With On-treatment Adverse Events (AES) and Serious Adverse Events(SAEs)
Description: An AE was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect. Data for on-treatment adverse events is reported.
Time Frame: Up to follow-up (5-10 days post last dose)
Population: All Subjects population.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Participants
  Any on-treatment AEs | 13 | 14 | 13 | 18
  Any on-treatment SAEs | 1 | 0 | 1 | 0

3. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure(DBP) at Specified Time Points in Semi-supine Position
Description: Blood pressure measurements were taken at pre-dose and at 120 min (completion of meal) on Day 1 and Day 28. The Baseline value was Day 1 Pre-Dose values. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 1, and Day 8
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Millimeters of mercury (mmHg)
  SBP Day 1 3.5 hours: number analyzed (Participants) | 13 | 13 | 13 | 15
  SBP Day 1 3.5 hours | 0.6 (13.68) | -1.8 (17.50) | 0.8 (18.07) | -2.3 (8.85)
  SBP Day 28 3.5 hours: number analyzed (Participants) | 11 | 13 | 13 | 15
  SBP Day 28 3.5 hours | 3.2 (12.09) | -1.1 (15.56) | 4.6 (16.47) | -7.2 (11.62)
  DBP Day 1 3.5 hours: number analyzed (Participants) | 13 | 13 | 13 | 15
  DBP Day 1 3.5 hours | -2.5 (8.09) | 1.1 (7.45) | -0.7 (8.50) | -2.3 (5.19)
  DBP Day 28 3.5 hours: number analyzed (Participants) | 11 | 13 | 13 | 15
  DBP Day 28 3.5 hours | -0.3 (4.69) | -0.8 (8.62) | 2.7 (6.33) | -6.1 (7.32)

4. Secondary Outcome: Change From Baseline in Heart Rate at Specified Time Points in Semi-supine Position
Description: Heart rate measurements were taken at pre-dose and 120 min (completion of meal) on Day 1 and Day 28. The Baseline value was Day 1 Pre-Dose values . Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 1, and Day 8
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Beats per minute (BPM)
  Heart rate Day 1 3.5 hours: number analyzed (Participants) | 13 | 13 | 13 | 15
  Heart rate Day 1 3.5 hours | -0.3 (7.60) | -0.8 (6.64) | -0.3 (8.39) | 2.1 (6.31)
  Heart rate Day 28 3.5 hours: number analyzed (Participants) | 11 | 13 | 13 | 15
  Heart rate Day 28 3.5 hours | -3.9 (6.86) | -1.5 (6.94) | 1.0 (9.09) | 0.7 (8.26)

5. Secondary Outcome: Change From Baseline in Electrocardiography Parameters (12-lead ECG)
Description: ECG measurements were taken at pre-dose and 0 min (completion of meal) on Day 1 and Day 28. The Baseline value was the Day 1 pre-dose value. ECG parameters included PR interval, QRS duration, QT interval, QTcB, QTcF and RR interval.
Time Frame: Baseline, Day 1 and Day 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Milliseconds (msec)
  PR interval Day 1 1.5 hours: number analyzed (Participants) | 19 | 18 | 17 | 22
  PR interval Day 1 1.5 hours | -2.6 (10.40) | 3.2 (7.46) | 0.5 (13.03) | -0.9 (9.68)
  PR interval Day 14 pre-dose: number analyzed (Participants) | 19 | 16 | 17 | 22
  PR interval Day 14 pre-dose | -5.5 (7.39) | 0.6 (7.87) | -1.6 (11.29) | -3.1 (9.25)
  PR interval Day 28 pre-dose: number analyzed (Participants) | 19 | 16 | 17 | 22
  PR interval Day 28 pre-dose | 2.4 (17.12) | -7.1 (26.93) | 2.2 (18.32) | -0.1 (8.14)
  PR interval Day 28 1.5 hours: number analyzed (Participants) | 18 | 15 | 17 | 21
  PR interval Day 28 1.5 hours | 1.2 (14.28) | 0.5 (11.48) | 3.6 (16.71) | -4.3 (9.54)
  QRS duration Day 1 1.5 hours | 0.2 (5.18) | -0.6 (4.16) | 0.1 (4.07) | 0.6 (5.22)
  QRS duration Day 14 pre-dose: number analyzed (Participants) | 20 | 16 | 18 | 22
  QRS duration Day 14 pre-dose | 0.1 (5.26) | -0.8 (4.33) | -0.1 (3.57) | -0.9 (4.97)
  QRS duration Day 28 pre-dose: number analyzed (Participants) | 19 | 16 | 18 | 22
  QRS duration Day 28 pre-dose | 2.4 (4.93) | 1.1 (4.54) | -0.3 (3.84) | 1.0 (4.81)
  QRS duration Day 28 1.5 hours: number analyzed (Participants) | 18 | 15 | 18 | 21
  QRS duration Day 28 1.5 hours | 0.8 (4.29) | 0.6 (3.98) | -0.3 (4.96) | 0.0 (4.97)
  QT interval Day 1 1.5 hours | 1.0 (12.30) | -0.2 (17.45) | -3.8 (13.16) | 1.6 (12.64)
  QT interval Day 14 pre-dose: number analyzed (Participants) | 20 | 16 | 18 | 22
  QT interval Day 14 pre-dose | -8.8 (18.52) | -9.6 (19.11) | -10.7 (25.58) | -9.6 (19.87)
  QT interval Day 28 pre-dose: number analyzed (Participants) | 19 | 16 | 18 | 22
  QT interval Day 28 pre-dose | 0.3 (21.83) | -5.0 (21.36) | -2.0 (23.20) | -3.0 (20.29)
  QT interval Day 28 1.5 hours: number analyzed (Participants) | 18 | 15 | 18 | 21
  QT interval Day 28 1.5 hours | 4.9 (16.37) | -2.8 (22.18) | -1.3 (26.49) | -4.5 (21.38)
  QTcB Day 1 1.5 hours: number analyzed (Participants) | 21 | 17 | 17 | 22
  QTcB Day 1 1.5 hours | -2.84 (13.906) | -1.94 (13.721) | -2.45 (13.447) | -0.12 (15.771)
  QTcB Day 14 pre-dose: number analyzed (Participants) | 20 | 15 | 17 | 22
  QTcB Day 14 pre-dose | 3.23 (11.503) | -2.97 (12.075) | -2.68 (18.410) | -1.42 (16.245)
  QTcB Day 28 pre-dose: number analyzed (Participants) | 19 | 15 | 17 | 22
  QTcB Day 28 pre-dose | -3.85 (20.907) | 2.71 (9.741) | 1.31 (18.419) | -0.20 (15.062)
  QTcB Day 28 1.5 hours: number analyzed (Participants) | 18 | 14 | 17 | 21
  QTcB Day 28 1.5 hours | 1.59 (24.246) | 1.86 (14.682) | -0.16 (17.208) | -0.88 (15.216)
  QTcF Day 1 1.5 hours: number analyzed (Participants) | 21 | 17 | 17 | 22
  QTcF Day 1 1.5 hours | -1.52 (12.089) | -1.26 (14.709) | -2.84 (11.080) | 0.72 (12.418)
  QTcF Day 14 pre-dose: number analyzed (Participants) | 20 | 15 | 17 | 22
  QTcF Day 14 pre-dose | -1.02 (11.942) | -5.57 (12.599) | -5.91 (19.109) | -4.37 (13.314)
  QTcF Day 28 pre-dose: number analyzed (Participants) | 19 | 15 | 17 | 22
  QTcF Day 28 pre-dose | -2.55 (18.782) | 0.04 (12.835) | 0.96 (15.942) | -1.21 (12.490)
  QTcF Day 28 1.5 hours: number analyzed (Participants) | 18 | 14 | 17 | 21
  QTcF Day 28 1.5 hours | 2.70 (20.473) | -0.24 (14.344) | -0.64 (16.857) | -2.17 (12.797)
  RR interval Day 1 1.5 hours: number analyzed (Participants) | 21 | 17 | 17 | 22
  RR interval Day 1 1.5 hours | 16.82 (56.084) | 7.26 (44.025) | -3.26 (68.824) | 8.74 (81.926)
  RR interval Day 14 pre-dose: number analyzed (Participants) | 20 | 15 | 17 | 22
  RR interval Day 14 pre-dose | -54.61 (76.965) | -33.95 (75.539) | -42.92 (90.333) | -35.25 (102.822)
  RR interval Day 28 pre-dose: number analyzed (Participants) | 19 | 15 | 17 | 22
  RR interval Day 28 pre-dose | 18.15 (109.227) | -31.14 (75.740) | -3.31 (99.049) | -11.51 (108.680)
  RR interval Day 28 1.5 hours: number analyzed (Participants) | 18 | 14 | 17 | 21
  RR interval Day 28 1.5 hours | 13.96 (76.906) | -23.69 (96.568) | -4.08 (114.019) | -15.60 (108.056)

6. Secondary Outcome: Number of Participants Outside the Normal Range for SBP and DBP
Description: Blood pressure measurements were taken at pre-dose and at 120 min (completion of meal) on Day 1 and Day 28. The clinical concern range (CCR) for SBP was greater than (<) 85 and less than (>) 160 and for DBP the range was <45 and >100. Data for semi-supine position has been presented. Baseline was Screening2/Baseline values.
Time Frame: Screening2/Baseline (Day -30 to -1), Day 1 and 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Participants
  SBP Screening 3.5 hours < CCR: number analyzed (Participants) | 13 | 13 | 13 | 15
  SBP Screening 3.5 hours < CCR | 0 | 0 | 0 | 0
  SBP Screening 3.5 hours>CCR: number analyzed (Participants) | 13 | 13 | 13 | 15
  SBP Screening 3.5 hours>CCR | 0 | 1 | 0 | 0
  SBP Day 1 3.5 hours< CCR: number analyzed (Participants) | 14 | 15 | 16 | 20
  SBP Day 1 3.5 hours< CCR | 0 | 0 | 1 | 0
  SBP Day 1 3.5 hours>CCR: number analyzed (Participants) | 14 | 15 | 16 | 20
  SBP Day 1 3.5 hours>CCR | 0 | 1 | 0 | 0
  SBP Day 28 3.5 hours< CCR: number analyzed (Participants) | 12 | 15 | 17 | 20
  SBP Day 28 3.5 hours< CCR | 0 | 0 | 0 | 0
  SBP Day 28 3.5 hours>CCR: number analyzed (Participants) | 12 | 15 | 17 | 20
  SBP Day 28 3.5 hours>CCR | 0 | 1 | 0 | 0
  DBP Screening 3.5 hours< CCR: number analyzed (Participants) | 13 | 13 | 13 | 15
  DBP Screening 3.5 hours< CCR | 0 | 0 | 0 | 0
  DBP Screening 3.5 hours>CCR: number analyzed (Participants) | 13 | 13 | 13 | 15
  DBP Screening 3.5 hours>CCR | 0 | 0 | 0 | 0
  DBP Day 1 3.5 hours: number analyzed (Participants) | 14 | 15 | 16 | 20
  DBP Day 1 3.5 hours | 0 | 0 | 0 | 0
  DBP Day 1 3.5 hours - 2 | 0 | 0 | 0 | 0
  DBP Day 28 3.5 hours: number analyzed (Participants) | 12 | 15 | 17 | 20
  DBP Day 28 3.5 hours | 0 | 0 | 0 | 0
  DBP Day 28 3.5 hours - 2 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Outside the Normal Range for Heart Rate
Description: Heart rate measurements were taken at pre-dose and at 120 min (completion of meal) on Day 1 and Day 28. The CCR for heart rate was Increase or decrease by less than or equal to (>=) 15 and >= 30. Data for semi-supine position has been presented. Baseline was Screening2/Baseline values.
Time Frame: Screening2/Baseline (Day -30 to -1), Day 1 and 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Participants
  Heart rate Screening 3.5 hours <CCR: number analyzed (Participants) | 13 | 13 | 13 | 15
  Heart rate Screening 3.5 hours <CCR | 0 | 0 | 0 | 0
  Heart rate Screening 3.5 hours >CCR: number analyzed (Participants) | 13 | 13 | 13 | 15
  Heart rate Screening 3.5 hours >CCR | 0 | 0 | 0 | 0
  Heart rate Day 1 3.5 hours <CCR: number analyzed (Participants) | 14 | 15 | 16 | 20
  Heart rate Day 1 3.5 hours <CCR | 0 | 0 | 0 | 0
  Heart rate Day 1 3.5 hours >CCR: number analyzed (Participants) | 14 | 15 | 16 | 20
  Heart rate Day 1 3.5 hours >CCR | 0 | 0 | 0 | 0
  Heart rate Day 28 3.5 hours<CCR: number analyzed (Participants) | 12 | 15 | 17 | 20
  Heart rate Day 28 3.5 hours<CCR | 0 | 0 | 0 | 0
  Heart rate Day 28 3.5 hours> CCR: number analyzed (Participants) | 12 | 15 | 17 | 20
  Heart rate Day 28 3.5 hours> CCR | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants Outside the Normal Range for 12-lead ECG
Description: ECG measurements were taken at pre-dose and 0 min (completion of meal) on Day 1 and Day 28. The CCR for ECG parameters were: PR interval (<110 and >220), QRS interval (<75 and >110), Absolute QTc interval (>450 to =< 480) respectively. Baseline was the pre-dose reading for Day 1. Data for abnormal- clinically significant (ACS) and abnormal- not clinically significant (ANCS) has been presented.
Time Frame: Baseline (Day 1 pre-dose), Day 1, Day 14 and Day 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Participants
  Day 1 pre-dose ANCS | 6 | 7 | 6 | 5
  Day 1 pre-dose ACS | 0 | 0 | 0 | 0
  Day 1 1.5 hour ANCS | 6 | 8 | 6 | 6
  Day 1 1.5 hour ACS | 0 | 0 | 0 | 0
  Day 14 pre-dose ANCS: number analyzed (Participants) | 20 | 16 | 18 | 22
  Day 14 pre-dose ANCS | 7 | 7 | 5 | 7
  Day 14 pre-dose ACS: number analyzed (Participants) | 20 | 16 | 18 | 22
  Day 14 pre-dose ACS | 0 | 0 | 0 | 0
  Day 28 pre-dose ANCS: number analyzed (Participants) | 19 | 16 | 18 | 22
  Day 28 pre-dose ANCS | 7 | 5 | 4 | 5
  Day 28 pre-dose ACS: number analyzed (Participants) | 19 | 16 | 18 | 22
  Day 28 pre-dose ACS | 0 | 0 | 0 | 0
  Day 28 1.5 hour ANCS: number analyzed (Participants) | 18 | 15 | 18 | 21
  Day 28 1.5 hour ANCS | 7 | 6 | 5 | 5
  Day 28 1.5 hour ACS: number analyzed (Participants) | 18 | 15 | 18 | 21
  Day 28 1.5 hour ACS | 0 | 0 | 0 | 0

9. Secondary Outcome: Mean Change From Baseline in Clinical Chemistry: Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, Gamma Glutamyl Transferase, Creatine Kinase, Lactate Dehydrogenase
Description: Alkaline phosphatase, alanine amino transferase, aspartate amino transferase, gamma glutamyl transferase, creatine kinase, lactate dehydrogenase measurements were taken at Baseline (Day 1 pre-dose), Day 5, 10, 14, 21 and 28. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Day 5, 10, 14, 21 and 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
International units per liter (IU/L)
  Alkaline Phosphatase Day 5: number analyzed (Participants) | 20 | 16 | 18 | 21
  Alkaline Phosphatase Day 5 | 3.0 (7.54) | 4.3 (7.20) | 4.0 (9.27) | -1.1 (23.56)
  Alkaline Phosphatase Day 10: number analyzed (Participants) | 19 | 16 | 18 | 21
  Alkaline Phosphatase Day 10 | 2.7 (8.63) | 5.0 (7.79) | 2.8 (10.58) | -1.3 (26.28)
  Alkaline Phosphatase Day 14: number analyzed (Participants) | 19 | 16 | 18 | 22
  Alkaline Phosphatase Day 14 | 3.7 (9.17) | 5.0 (8.16) | 0.7 (8.70) | -4.3 (24.67)
  Alkaline Phosphatase Day 21: number analyzed (Participants) | 18 | 16 | 18 | 22
  Alkaline Phosphatase Day 21 | 4.3 (15.25) | 3.9 (9.19) | 1.7 (11.39) | -1.7 (26.96)
  Alkaline Phosphatase Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Alkaline Phosphatase Day 28 | 1.1 (14.05) | 3.1 (7.17) | -2.5 (14.66) | -1.7 (25.23)
  Alanine Amino Transferase Day 5: number analyzed (Participants) | 20 | 16 | 18 | 21
  Alanine Amino Transferase Day 5 | 0.7 (3.28) | 2.6 (7.31) | 2.8 (10.88) | -1.1 (16.03)
  Alanine Amino Transferase Day 10: number analyzed (Participants) | 19 | 16 | 18 | 21
  Alanine Amino Transferase Day 10 | 0.6 (7.86) | 2.5 (6.60) | -1.2 (4.93) | -1.1 (17.05)
  Alanine Amino Transferase Day 14: number analyzed (Participants) | 19 | 16 | 18 | 22
  Alanine Amino Transferase Day 14 | 2.4 (7.32) | 2.9 (6.99) | -1.0 (6.94) | -3.2 (15.94)
  Alanine Amino Transferase Day 21: number analyzed (Participants) | 18 | 16 | 18 | 22
  Alanine Amino Transferase Day 21 | -0.4 (6.74) | 0.3 (6.09) | -0.1 (5.89) | -2.9 (14.59)
  Alanine Amino Transferase Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Alanine Amino Transferase Day 28 | -1.5 (5.39) | 1.1 (6.22) | -1.2 (6.88) | -4.0 (13.60)
  Aspartate Amino Transferase Day 5 | -0.3 (5.68) | 0.1 (6.73) | -1.9 (9.90) | 1.6 (4.56)
  Aspartate Amino Transferase Day 10: number analyzed (Participants) | 19 | 16 | 18 | 21
  Aspartate Amino Transferase Day 10 | 0.5 (9.08) | 1.2 (8.27) | -2.7 (10.67) | 2.8 (3.43)
  Aspartate Amino Transferase Day 14: number analyzed (Participants) | 19 | 16 | 18 | 22
  Aspartate Amino Transferase Day 14 | 2.6 (5.50) | -1.1 (6.94) | -2.8 (11.35) | 1.0 (6.36)
  Aspartate Amino Transferase Day 21: number analyzed (Participants) | 18 | 16 | 18 | 22
  Aspartate Amino Transferase Day 21 | -1.1 (6.80) | -0.3 (6.78) | -1.2 (9.55) | 1.6 (5.12)
  Aspartate Amino Transferase Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Aspartate Amino Transferase Day 28 | -0.8 (6.63) | 0.4 (5.41) | -2.7 (9.13) | 0.5 (6.61)
  Gamma Glutamyl Transferase Day 5: number analyzed (Participants) | 20 | 14 | 13 | 18
  Gamma Glutamyl Transferase Day 5 | -0.5 (2.43) | 1.8 (4.35) | 1.6 (6.26) | 2.4 (8.44)
  Gamma Glutamyl Transferase Day 10: number analyzed (Participants) | 18 | 15 | 13 | 20
  Gamma Glutamyl Transferase Day 10 | -1.1 (2.88) | 0.5 (4.16) | 1.8 (7.09) | 1.2 (6.79)
  Gamma Glutamyl Transferase Day 14: number analyzed (Participants) | 20 | 14 | 16 | 20
  Gamma Glutamyl Transferase Day 14 | -0.2 (4.57) | 0.4 (3.10) | 2.1 (6.55) | 1.5 (8.95)
  Gamma Glutamyl Transferase Day 21: number analyzed (Participants) | 17 | 15 | 14 | 20
  Gamma Glutamyl Transferase Day 21 | -0.3 (5.11) | -1.3 (5.00) | 1.8 (3.52) | 2.6 (7.93)
  Gamma Glutamyl Transferase Day 28: number analyzed (Participants) | 19 | 15 | 17 | 21
  Gamma Glutamyl Transferase Day 28 | -1.7 (5.44) | 0.5 (5.51) | 0.3 (4.37) | 4.2 (16.01)
  Creatine Kinase Day 28: number analyzed (Participants) | 17 | 11 | 11 | 17
  Creatine Kinase Day 28 | -4.3 (61.05) | 41.9 (74.29) | 42.0 (103.49) | 0.2 (42.14)
  Lactate Dehydrogenase Day 28: number analyzed (Participants) | 16 | 12 | 12 | 17
  Lactate Dehydrogenase Day 28 | -11.5 (38.69) | 8.6 (31.10) | -5.8 (42.29) | -16.2 (40.37)

10. Secondary Outcome: Mean Change From Baseline in Clinical Chemistry: Direct Bilirubin, Total Bilirubin, Creatinine, Uric Acid
Description: Direct Bilirubin, Total Bilirubin, Creatinine, Uric acid measurements were taken at Baseline (Day 1 pre-dose), Day 5, 10, 14, 21 and 28. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline (Day 1 pre-dose), Day 5, 10, 14, 21 and 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Unit moles per litre (UMOL/L)
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Unit moles per litre (UMOL/L)
  Direct Bilirubin Day 5: number analyzed (Participants) | 20 | 15 | 14 | 19
  Direct Bilirubin Day 5 | 0.1 (0.75) | -0.2 (1.27) | -0.1 (0.62) | -0.0 (1.38)
  Direct Bilirubin Day 10: number analyzed (Participants) | 19 | 13 | 14 | 19
  Direct Bilirubin Day 10 | 0.1 (0.75) | 0.0 (1.65) | -0.1 (0.75) | -0.0 (1.10)
  Direct Bilirubin Day 14: number analyzed (Participants) | 20 | 14 | 14 | 20
  Direct Bilirubin Day 14 | 0.1 (0.57) | 0.1 (1.19) | -0.2 (0.70) | -0.0 (1.21)
  Direct Bilirubin Day 21: number analyzed (Participants) | 17 | 14 | 14 | 20
  Direct Bilirubin Day 21 | 0.1 (0.75) | 0.2 (1.35) | -0.2 (0.90) | 0.1 (1.03)
  Direct Bilirubin Day 28: number analyzed (Participants) | 19 | 14 | 14 | 19
  Direct Bilirubin Day 28 | 0.1 (0.74) | 0.3 (1.57) | 0.1 (0.98) | -0.1 (0.84)
  Total Bilirubin Day 5: number analyzed (Participants) | 20 | 16 | 18 | 21
  Total Bilirubin Day 5 | 0.2 (2.43) | 0.4 (2.71) | -2.6 (3.41) | -0.5 (3.19)
  Total Bilirubin Day 10: number analyzed (Participants) | 19 | 16 | 18 | 21
  Total Bilirubin Day 10 | -0.4 (2.25) | -0.1 (3.13) | -1.8 (4.83) | -0.4 (2.57)
  Total Bilirubin Day 14: number analyzed (Participants) | 19 | 16 | 18 | 22
  Total Bilirubin Day 14 | 0.5 (2.41) | 0.2 (2.99) | -2.1 (3.15) | -0.3 (2.99)
  Total Bilirubin Day 21: number analyzed (Participants) | 18 | 16 | 18 | 22
  Total Bilirubin Day 21 | -0.6 (2.53) | 0.4 (3.72) | -1.2 (3.49) | -0.2 (1.99)
  Total Bilirubin, Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Total Bilirubin, Day 28 | 0.0 (1.87) | 1.2 (3.45) | -0.6 (2.71) | -0.9 (3.27)
  Creatinine Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Creatinine Day 28 | -2.91 (6.156) | 0.51 (7.415) | 9.42 (17.103) | 9.80 (11.993)
  Uric acid Day 28: number analyzed (Participants) | 19 | 15 | 17 | 22
  Uric acid Day 28 | -8.61 (39.359) | 3.56 (32.183) | 8.62 (25.412) | 18.29 (39.987)

11. Secondary Outcome: Mean Change From Baseline in Clinical Chemistry : Albumin, Total Protein
Description: Albumin, Total Protein measurements were taken at Baseline (Day 1 pre-dose), and Day 28. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Grams per liter (g/L)
  Albumin Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Albumin Day 28 | -0.68 (2.335) | 0.49 (2.040) | 0.11 (1.323) | -0.66 (2.308)
  Total Protein Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Total Protein Day 28 | -0.3 (3.79) | 0.7 (2.94) | 1.0 (2.68) | -0.5 (4.53)

12. Secondary Outcome: Mean Change From Baseline in Clinical Chemistry : Calcium, Chloride, Glucose, Potassium, Sodium, Urea/BUN, Carbon Dioxide Content/Bicarbonate
Description: Calcium, Chloride, Glucose, Potassium, Sodium, Urea/BUN, Carbon dioxide content/Bicarbonate measurements were taken at Baseline (Day 1 pre-dose) and Day 28. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (MMOL/L)
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Millimoles per liter (MMOL/L)
  Calcium Day 28: number analyzed (Participants) | 19 | 16 | 17 | 22
  Calcium Day 28 | -0.018 (0.1067) | -0.017 (0.0764) | 0.027 (0.0666) | -0.031 (0.1323)
  Chloride Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Chloride Day 28 | 0.26 (3.754) | -0.93 (3.137) | -0.94 (2.578) | 0.15 (2.759)
  Glucose Day 28: number analyzed (Participants) | 18 | 16 | 18 | 22
  Glucose Day 28 | -0.21 (4.343) | 0.24 (3.638) | 0.66 (6.790) | -0.25 (2.332)
  Potassium Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Potassium Day 28 | -0.042 (0.3564) | 0.094 (0.6002) | -0.111 (0.5132) | -0.068 (0.3999)
  Sodium Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Sodium Day 28 | -0.42 (3.203) | -0.41 (2.303) | -0.56 (2.833) | 0.00 (1.718)
  Urea/BUN Day 28: number analyzed (Participants) | 17 | 12 | 15 | 19
  Urea/BUN Day 28 | -0.35 (2.021) | -0.31 (1.778) | -0.04 (1.942) | 0.26 (2.016)
  Carbon dioxide content/Bicarbonate Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Carbon dioxide content/Bicarbonate Day 28 | -0.21 (1.843) | -0.79 (2.286) | 1.17 (2.526) | -0.08 (2.298)

13. Secondary Outcome: Mean Change From Baseline in Hematology Parameters : Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils (Total ANC - Total Absolute Neutrophil Count), Platelet Count, White Blood Cell Count
Description: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils (Total ANC - Total Absolute Neutrophil Count), Platelet count, White Blood cell count measurements were taken at Baseline (Day 1 pre-dose) and Day 28. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells per liter (GI/L)
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Giga (10^9) cells per liter (GI/L)
  Basophils Day 28: number analyzed (Participants) | 19 | 16 | 16 | 21
  Basophils Day 28 | 0.0066 (0.03852) | -0.0388 (0.09539) | -0.0322 (0.07998) | 0.1072 (0.43592)
  Eosinophils Day 28: number analyzed (Participants) | 19 | 16 | 17 | 21
  Eosinophils Day 28 | -0.0167 (0.07137) | 0.0431 (0.11412) | -0.0040 (0.18975) | 0.1173 (0.41877)
  Lymphocytes Day 28: number analyzed (Participants) | 19 | 16 | 18 | 21
  Lymphocytes Day 28 | 0.0485 (0.44972) | -0.0561 (0.45151) | 0.1887 (0.31662) | -0.0099 (0.34075)
  Monocytes Day 28: number analyzed (Participants) | 19 | 16 | 18 | 21
  Monocytes Day 28 | -0.0327 (0.16668) | -0.0530 (0.09965) | -0.0097 (0.17272) | -0.0298 (0.10623)
  Total Neutrophils Day 28: number analyzed (Participants) | 19 | 16 | 18 | 21
  Total Neutrophils Day 28 | 0.1380 (0.78256) | 0.2159 (1.28307) | 0.2949 (1.20093) | -0.7640 (1.97899)
  Platelet count Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Platelet count Day 28 | 6.4 (32.76) | 1.5 (35.37) | 0.6 (28.87) | -2.0 (21.58)
  White Blood cell count Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  White Blood cell count Day 28 | 0.144 (1.0951) | 0.225 (1.4369) | 0.428 (1.0110) | -0.730 (2.0794)

14. Secondary Outcome: Mean Change From Baseline in Hematology Parameters : Hematocrit
Description: Hematocrit measurements were taken at Baseline (Day 1 pre-dose) and Day 28. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 19 | 16 | 18 | 22
Ratio | -0.0025 (0.01692) | 0.0021 (0.01053) | 0.0019 (0.01508) | -0.0059 (0.01637)

15. Secondary Outcome: Mean Change From Baseline in Hematology Parameters : Mean Corpuscle Hemoglobin
Description: Mean Corpuscle Hemoglobin measurements were taken at Baseline (Day 1 pre-dose) and Day 28. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms (Pg)
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 17 | 14 | 15 | 19
Picograms (Pg) | 0.05 (0.521) | 0.15 (0.454) | -0.15 (0.667) | -0.14 (0.643)

16. Secondary Outcome: Mean Change From Baseline in Hematology Parameters : Hemoglobin, Mean Corpuscle Hemoglobin Concentration
Description: Hemoglobin, Mean Corpuscle Hemoglobin concentration measurements were taken at Baseline (Day 1 pre-dose) and Day 28. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
g/L
  Hemoglobin Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Hemoglobin Day 28 | 0.4 (5.36) | 1.1 (4.63) | -0.2 (5.46) | -2.7 (5.11)
  Mean Corpuscle Hemoglobin concentration Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Mean Corpuscle Hemoglobin concentration Day 28 | 2.8 (6.20) | 1.6 (4.92) | -2.8 (6.53) | -1.9 (7.81)

17. Secondary Outcome: Mean Change From Baseline in Hematology Parameters : Mean Corpuscle Volume
Description: Mean Corpuscle Volume measurements were taken at Baseline (Day 1 pre-dose) and Day 28. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters (FL)
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 19 | 16 | 18 | 22
Femtoliters (FL) | -0.52 (0.952) | -0.24 (1.163) | 0.43 (1.514) | 0.13 (1.318)

18. Secondary Outcome: Mean Change From Baseline in Hematology Parameters : Red Blood Cell Count, Reticulocytes
Description: Red Blood Cell count, Reticulocytes measurements were taken at Baseline (Day 1 pre-dose) and Day 28. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Tera (10^12) cells per liter (TI/L)
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Tera (10^12) cells per liter (TI/L)
  Red Blood Cell count Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Red Blood Cell count Day 28 | 0.003 (0.2015) | 0.035 (0.1399) | 0.003 (0.1597) | -0.072 (0.1660)
  Reticulocytes Day 28: number analyzed (Participants) | 19 | 16 | 18 | 22
  Reticulocytes Day 28 | -0.0080 (0.02949) | -0.0051 (0.01418) | 0.0070 (0.01919) | -0.0050 (0.01937)

19. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration AUC(0-t) at Specified Time Points
Description: AUC(0-t) was derived from GSK962040 plasma concentration-time data. AUC was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.Only participants who received GSK962040 drug were analyzed.
Time Frame: Pre-dose and 1.5, 2.5, 3.5, 4.5, and 5.5 hours post dose on Day 1 and 28
Population: The 'Pharmacokinetic (PK) Population' was defined as participants in the 'All subjects' population for whom a PK sample was obtained and analyzed. Only those participants available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms.hour/milliliter (ng.h/mL)
Arm/Group | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 18 | 18 | 22
Nanograms.hour/milliliter (ng.h/mL)
  Day 1: number analyzed (Participants) | 15 | 18 | 21
  Day 1 | 854.9 (36.6) | 4083.1 (23.6) | 12911.9 (30.0)
  Day 28: number analyzed (Participants) | 15 | 15 | 21
  Day 28 | 1908.1 (46.1) | 7347.2 (24.3) | 22173.3 (31.8)

20. Secondary Outcome: Maximum Observed Concentration (Cmax) at Specified Time Points
Description: Cmax is defined as the maximum observed drug concentration after administration. Cmax was determined directly from the raw concentration-time data. Samples were collected at the following times: Pre-dose and 1.5, 2.5, 3.5, 4.5, and 5.5 hours post dose.
Time Frame: Pre-dose and 1.5, 2.5, 3.5, 4.5, and 5.5 hours post dose on Day 1 and 28
Population: PK population. Only those participants available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 18 | 18 | 22
Nanograms per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 15 | 18 | 21
  Day 1 | 70.21 (54.7) | 385.73 (27.6) | 1239.62 (40.0)
  Day 28: number analyzed (Participants) | 15 | 15 | 21
  Day 28 | 131.71 (52.9) | 530.97 (34.0) | 1703.29 (38.0)

21. Secondary Outcome: Time of Occurrence of Cmax (Tmax) at Specified Time Points
Description: Tmax is defined as the time to reach the observed maximum concentration. Samples were collected at the following times: Tmax was determined directly from the raw concentration-time data. Pre-dose and 1.5, 2.5, 3.5, 4.5, and 5.5 hours post dose.
Time Frame: Pre-dose and 1.5, 2.5, 3.5, 4.5, and 5.5 hours post dose on Day 1 and 28
Population: PK population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 18 | 18 | 22
Hour
  Day 1: number analyzed (Participants) | 15 | 18 | 21
  Day 1 | 2.174 (0.9066) | 2.238 (1.0697) | 2.092 (0.8419)
  Day 28: number analyzed (Participants) | 15 | 15 | 21
  Day 28 | 2.189 (1.3976) | 2.168 (0.7224) | 2.026 (1.2038)

22. Secondary Outcome: Pre-dose (Trough) Concentration at the End of the Dosing Interval (Ct) at Specified Time Points
Description: Analysis of pre-dose (trough) concentration at the end of the dosing interval (Ct) was planned to be performed from the samples collected at Pre -dose and 1.5, 2.5, 3.5, 4.5, and 5.5 hours post dose on Day 1 and 28.
Time Frame: Pre-dose and 1.5, 2.5, 3.5, 4.5, and 5.5 hours post dose on Day 1 and 28
Population: PK population.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 18 | 18 | 22
Liters
  Day 14: number analyzed (Participants) | 14 | 18 | 21
  Day 14 | 63.73 (34.853) | 214.26 (146.572) | 537.23 (290.370)
  Day 28: number analyzed (Participants) | 15 | 15 | 21
  Day 28 | 62.60 (32.830) | 205.03 (84.251) | 597.39 (321.225)

23. Secondary Outcome: Apparent Clearance Following Oral Dosing (CL/F) at Specified Time Points
Description: CL/F was calculated as dose/AUC. The parameter was planned to be analyzed from samples collected at Pre -dose and 1.5, 2.5, 3.5, 4.5, and 5.5 hours post dose on Day 1 and 28, however the data for this outcome measure was not collected.
Time Frame: Pre-dose and 1.5, 2.5, 3.5, 4.5, and 5.5 hours post dose on Day 1 and 28
Population: PK Population. The data for this outcome measure was not collected.
Arm/Group | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Apparent Volume of Distribution (V/F) at Specified Time Points
Description: The apparent volume of distribution V/F = CL/F × MRT, where MRT is the mean residence time. The parameter was planned to be analyzed using samples collected at Pre-dose and 1.5, 2.5, 3.5, 4.5, and 5.5 hours post dose on Day 1 and 28, however, the data for this outcome measure was not collected.
Time Frame: Pre-dose and 1.5, 2.5, 3.5, 4.5, and 5.5 hours post dose on Day 1 and 28
Population: PK Population. The data for this outcome measure was not collected.
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

25. Secondary Outcome: Apparent Terminal Elimination Half-life (t1/2) at Specified Time Points
Description: This outcome measure was not analyzed in results.
Time Frame: The parameter was planned to be analyzed using samples collected at Pre-dose and 1.5, 2.5, 3.5, 4.5, and 5.5 hours post dose on Day 1 and 28, however, the data for this outcome measure was not collected.
Population: PK Population. The data for this outcome measure was not collected.
Arm/Group | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 0 | 0 | 0

26. Secondary Outcome: Time to First Bowel Movement After First Dose
Description: The time to first bowel movement was calculated as the time of the first bowel movement after the first dose in hours (floored) for each participant. If a participant had fewer than 5 days worth of data then the daily mean for that week was set to missing for the following two parameters: Bowel Movement Count and Stool Consistency. Seventeen participants who entered their time of first instance of bowel movement before taking first dose were excluded from the summary statistics of time to first bowel movement.
Time Frame: Up to Day 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 16 | 12 | 15 | 12
hours | 28.94 (25.044) | 53.98 (67.901) | 17.52 (19.286) | 15.73 (15.648)

27. Secondary Outcome: Daily Bowel Movement Frequency
Description: Daily bowel movement frequency analyzed number of times passed stools in 24 hours of duration. Following dosing with study medication, stool monitoring was performed up to Day 28. Seventeen participants who entered their time of first instance of bowel movement before taking first dose were excluded from the summary statistics.
Time Frame: Up to Week 4 (Day 28)
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Bowel movements/24 hours
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Bowel movements/24 hours
  Week 1: number analyzed (Participants) | 19 | 11 | 17 | 21
  Week 1 | 1.30 (0.872) | 1.33 (0.812) | 1.50 (0.943) | 1.39 (0.729)
  Week 2: number analyzed (Participants) | 20 | 14 | 17 | 22
  Week 2 | 2.23 (3.473) | 1.59 (0.948) | 1.55 (1.012) | 1.45 (0.883)
  Week 3: number analyzed (Participants) | 19 | 15 | 17 | 22
  Week 3 | 2.18 (3.269) | 1.44 (0.830) | 1.77 (1.172) | 1.38 (0.770)
  Week 4: number analyzed (Participants) | 17 | 16 | 17 | 21
  Week 4 | 2.11 (3.432) | 1.54 (0.841) | 1.68 (1.049) | 1.37 (0.831)

28. Secondary Outcome: Daily Average Stool Consistency
Description: Stool consistency was determined on a scale of 1 to 5 (1 = Very hard, 2 = Hard, 3 = Formed, 4 = Loose, 5 = Watery). Following dosing with study medication, stool monitoring was performed up to Day 28. Participants who entered their time of first instance of bowel movement before taking first dose were excluded from the summary statistics.
Time Frame: Up to Week 4 (Day 28)
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Bowel Movements/ 24 hours
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Bowel Movements/ 24 hours
  Week 1: number analyzed (Participants) | 9 | 7 | 11 | 13
  Week 1 | 2.91 (0.817) | 3.24 (0.524) | 2.80 (0.815) | 3.71 (0.874)
  Week 2: number analyzed (Participants) | 13 | 11 | 13 | 17
  Week 2 | 2.98 (0.730) | 2.81 (0.673) | 3.05 (0.798) | 3.29 (0.724)
  Week 3: number analyzed (Participants) | 14 | 12 | 12 | 16
  Week 3 | 2.89 (0.517) | 2.87 (0.889) | 2.99 (0.558) | 3.26 (0.683)
  Week 4: number analyzed (Participants) | 12 | 13 | 12 | 14
  Week 4 | 2.92 (0.528) | 2.96 (0.625) | 2.98 (0.502) | 3.37 (0.569)

29. Secondary Outcome: Change From Baseline in Upper Gastrointestinal (GI) Symptoms as Assessed by Total Gastrointestinal Cardinal Symptom Index - Daily Diary (GCSI-DD)
Description: GCSI-DD was measured on a 6-point scale. The Total GCSI-DD score was the mean of the following three subscales: Nausea/Vomiting Subscale = mean (nausea, retching, vomiting), Fullness/Early Satiety Subscale = mean (feeling excessively full after meals, not able to finish a normal-sized meal, stomach fullness, loss of appetite), Bloating Subscale = mean (bloating, stomach or belly visibly larger). Each subscale was scored on a severity scale of 0 (none) to 5 (very severe), with lower scores representing less symptom severity. The change from Baseline to each study week in average score was derived and if it improved by 1 point or more, that participant was defined as "responder" for that symptom and on that particular week. Baseline was Screening2/Baseline values (Day -30 to -1). Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Up to 14 days post last dose (Day 28)
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
Score on a scale
  Week 1: number analyzed (Participants) | 19 | 11 | 17 | 21
  Week 1 | -0.48 (0.645) | -0.46 (0.676) | -0.58 (0.379) | -0.57 (0.491)
  Week 2: number analyzed (Participants) | 20 | 14 | 17 | 22
  Week 2 | -0.68 (0.728) | -1.04 (1.062) | -1.21 (0.663) | -0.72 (0.597)
  Week 3: number analyzed (Participants) | 19 | 15 | 17 | 22
  Week 3 | -0.75 (0.770) | -1.29 (0.936) | -1.16 (0.745) | -0.77 (0.654)
  Week 4: number analyzed (Participants) | 16 | 16 | 16 | 22
  Week 4 | -0.86 (1.001) | -1.32 (0.980) | -1.12 (0.670) | -0.82 (0.727)
  Week 5: number analyzed (Participants) | 18 | 15 | 16 | 22
  Week 5 | -0.87 (0.951) | -1.19 (0.906) | -1.07 (0.738) | -0.74 (0.728)
  Week 6: number analyzed (Participants) | 17 | 13 | 14 | 21
  Week 6 | -0.85 (0.943) | -0.96 (1.000) | -0.86 (0.632) | -0.59 (0.776)

30. Secondary Outcome: Change From Baseline in Whole Bowel Transit Time, 100 % Gastric Emptying Time (Truncated at 240 Minutes), Small Bowel Transit Time, Colonic Transit Time as Determined by Wireless Motility Capsule (WMC)
Description: WMC is an ingestible telemetric capsule which measures pH, pressure and temperature to assess total gastric emptying time, small and large bowel transit time, colonic transit time, and whole gut transit time. The WMC was ingested immediately following the standard test meal for the oral breath test. Data was collected on a data logger, which was worn on a belt clip. The WMC passed naturally in the participant's stools between 2 and 5 days after ingestion. The parameters Whole bowel transit time, 100 % gastric emptying time (truncated at 240 minutes), small bowel transit time, colonic transit time were analyzed. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline(Screening i.e., Day -30 to -1), Day 1 and 28
Population: All Subjects Population. Only those participants available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
Number analyzed (Participants) | 21 | 18 | 18 | 22
minutes
  100% Gastric Emptying Time Day 1: number analyzed (Participants) | 16 | 15 | 16 | 22
  100% Gastric Emptying Time Day 1 | -159.9 (616.67) | -240.3 (567.18) | -323.8 (461.05) | -381.0 (541.73)
  100% Gastric Emptying Time Day 28: number analyzed (Participants) | 14 | 14 | 14 | 22
  100% Gastric Emptying Time Day 28 | -243.0 (500.49) | -15.4 (502.80) | -162.7 (558.96) | -341.3 (599.52)
  100% Gastric Emptying Time(Truncated) Day 1: number analyzed (Participants) | 16 | 15 | 16 | 22
  100% Gastric Emptying Time(Truncated) Day 1 | 2.7 (27.95) | 3.7 (28.87) | -15.8 (61.32) | -65.5 (91.11)
  100% Gastric Emptying Time(Truncated) Day 28: number analyzed (Participants) | 14 | 14 | 14 | 22
  100% Gastric Emptying Time(Truncated) Day 28 | -10.7 (18.60) | 19.7 (42.47) | -13.9 (42.34) | -40.2 (68.66)
  Colonic Transit Time Day 1: number analyzed (Participants) | 16 | 14 | 15 | 21
  Colonic Transit Time Day 1 | -331.3 (1349.11) | -92.9 (1970.38) | -170.5 (1723.01) | -598.3 (1617.05)
  Colonic Transit Time Day 28: number analyzed (Participants) | 14 | 12 | 14 | 21
  Colonic Transit Time Day 28 | -518.1 (2650.06) | 142.9 (1326.20) | -29.4 (1702.69) | -416.4 (1447.79)
  Small Bowel Transit Time Day 1: number analyzed (Participants) | 16 | 14 | 15 | 21
  Small Bowel Transit Time Day 1 | -24.5 (118.39) | -47.7 (94.33) | 15.7 (211.88) | -6.6 (149.11)
  Small Bowel Transit Time 28: number analyzed (Participants) | 14 | 12 | 14 | 21
  Small Bowel Transit Time 28 | -76.4 (107.89) | -57.3 (176.42) | -7.1 (148.51) | -28.6 (135.44)
  Whole Bowel Transit Time Day 1: number analyzed (Participants) | 16 | 14 | 15 | 21
  Whole Bowel Transit Time Day 1 | -527.6 (1489.02) | -402.1 (2109.06) | -493.1 (1987.51) | -1002.5 (2045.60)
  Whole Bowel Transit Time 28: number analyzed (Participants) | 16 | 12 | 15 | 21
  Whole Bowel Transit Time 28 | -777.6 (2644.80) | -2.4 (1298.37) | -233.5 (1850.91) | -789.1 (1560.06)

ADVERSE EVENTS:
Time Frame: Up to follow-up i.e., 14 days ± 2 days post last dose (Day 28)
Description: All Subjects population was used to assess adverse events.
Arm/Group | Placebo | GSK962040 10 mg | GSK962040 50 mg | GSK962040 125 mg
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/18 | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/18 | 1/18 | 0/22
Other Adverse Events (participants affected / at risk) | 11/21 | 14/18 | 14/18 | 14/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | GSK962040 10 mg (N=18) | GSK962040 50 mg (N=18) | GSK962040 125 mg (N=22)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | GSK962040 10 mg (N=18) | GSK962040 50 mg (N=18) | GSK962040 125 mg (N=22)
Headache (Nervous system disorders) | 4 (5) | 2 (3) | 4 (6) | 6 (9)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 4 (5) | 3 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2) | 4 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (3) | 0 (0) | 1 (1) | 2 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (2) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 3 (4) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Feeling of body temperature change (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Energy increased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Painful defaecation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.